CLINICAL TRIAL: NCT03559426
Title: Research Into Antipsychotic Discontinuation and Reduction (RADAR): A Randomised Controlled Trial
Brief Title: Research Into Antipsychotic Discontinuation and Reduction Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/0947
Record Dates: First submitted 2018-05-29; First posted 2018-06-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder; Schizophreniform Disorders
Keywords: antipsychotics; schizophrenia; reduction
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid

STUDY DESIGN:
Intervention Model Description: Open, parallel group, multi-centre randomised controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Participants and treating clinicians will not be blinded because participants will start on different antipsychotic regimes, and those within the antipsychotic reduction intervention will follow an individualised reduction protocol.
  Following trial extension the sample size was reduced from 402 to 218. The study is now powered to the primary outcome 'social functioning'.
  Members of the research team conducting outcome assessments will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Antipsychotic Maintenance (Active Comparator): Participants continue to receive antipsychotic treatment at the original dose for the 24 month duration of the trial. Increases or minor adjustments to antipsychotic medication are permitted.
  Interventions: Drug: Antipsychotic Maintenance
- Antipsychotic Reduction (Experimental): Antipsychotic medication is gradually reduced and discontinued if possible. A flexible individualised antipsychotic reduction schedule is devised for each patient by the research team, based on the participant's initial antipsychotic regime. Antipsychotic dose is reduced incrementally every two months, with flexibility to speed up or slow down the schedule in discussion with the patient. The antipsychotic reduction extends over a period of between six to 12 months, although this may be extended according to individual circumstances.
  Interventions: Drug: Antipsychotic Reduction

INTERVENTIONS:
Drug: Antipsychotic Reduction — Antipsychotic medication is gradually reduced and discontinued if possible. A flexible individualised antipsychotic reduction schedule is devised for each patient by the research team, based on the participant's initial antipsychotic regime. Antipsychotic dose is reduced incrementally every two months, with flexibility to speed up or slow down the schedule in discussion with the patient. The antipsychotic reduction extends over a period of between six to 12 months, although this may be extended according to individual circumstances.
  Arms: Antipsychotic Reduction
Drug: Antipsychotic Maintenance — Participants continue to receive antipsychotic treatment at the original dose for the 24 month duration of the trial. Increases or minor adjustments to antipsychotic medication are permitted.
  Arms: Antipsychotic Maintenance

SUMMARY:
Psychosis and schizophrenia are common and costly mental health problems. Psychosis is the name given to a group of mental conditions in which cause people to perceive or interpret things differently from those around them. One of the most common causes of psychosis is schizophrenia, a condition that causes a range of psychological symptoms, including hallucinations (hearing and/or seeing things) and delusions (believing something that is not true). One of the main treatment options for psychosis and schizophrenia is long-term treatment with antipsychotic medication, but many patients still find life difficult. Antipsychotic drugs can also have dangerous and unpleasant side effects. Finding alternatives to long-term drug treatment is a priority for patients and services. This study is testing the effects of gradually reducing antipsychotic medication in people with schizophrenia, psychosis or similar conditions in order to see if it can help improve day-to-day functioning and how it affects their chance of suffering a relapse (worsening of their condition).

DETAILED DESCRIPTION:
The RADAR trial is a randomised controlled trial that will compare a flexible and gradual strategy of antipsychotic reduction and possible discontinuation with maintenance antipsychotic treatment in people with schizophrenia or who have recurrent psychotic episodes. In the reduction group, a guideline reduction schedule will be devised by the research team for each participant taking into account starting dose and number of antipsychotics prescribed. This may be adjusted by treating clinicians in discussion with participants. Antipsychotics will be discontinued in cases where reduction progresses well. The reduction schedule will be flexible, and will include guidance on monitoring and treating symptoms and signs of early relapse.

Participants will be individually randomised to the two treatment strategies, which will be administered by treating clinicians. They will be followed up for two years. The primary outcome is social functioning, and secondary outcomes include relapse, symptoms, side effects, employment and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* A clinical and/or ICD10 diagnosis of schizophrenia, schizoaffective disorder, delusional disorder or other non-affective psychosis
* More than one previous episode of relapse or psychotic exacerbation, or a single episode lasting more than one year
* Taking antipsychotic medication

Exclusion Criteria:

* Participant lacks capacity to consent to the trial
* Participant has insufficient command of spoken English to understand trial procedures
* Participant subject to section 37/41 of the Mental Health Act (MHA) or a Community Treatment Order (CTO) that includes a requirement to take antipsychotic medication.
* Clinician considers there will be a serious risk of harm to self or others
* Participant has been admitted to hospital or had treatment from the Home Treatment or Crisis Team within the last month
* Females who have a confirmed pregnancy
* Females who are breast-feeding
* Involvement in another "investigational medicinal product" (IMP) trial
* No contraindications to continuing on antipsychotic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Social Functioning Scale (Assessing change over time) | Baseline, 6 months, 12 months, 24 months
  Evaluates how the patient functions in daily living and social skills

SECONDARY OUTCOMES:
Severe relapse | Duration of the trial follow-up (24 months)
  Severe relapse is defined as admission to hospital for a relapse of a psychotic condition.
Positive and Negative Syndrome Scale (PANSS) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Clinical assessment of current symptomology. Measure refers to prevalence of psychotic symptoms ranging from absent to extreme.
Modified Glasgow Antipsychotics Side-Effects Scale (GASS) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Self-report measure of physical and mental side effects patient has experienced recently. Scale refers to prevalence of side effects from antipsychotic medication in the last week.
Manchester Short Assessment of Quality of Life (MANSA) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Assessment of quality of life.
Digit Span (forwards and backwards) Assessing change over time | Baseline,12 months, 24 months
  Neuropsychological assessment of short-term memory and attention
Digit Symbol Coding (Assessing change over time) | Baseline,12 months, 24 months
  A neuropsychological assessment of motor skill and attention
Rey Auditory Verbal Learning (Assessing change over time) | Baseline,12 months, 24 months
  Neuropsychological assessment of short-term memory and learning
Trail Making Test (Assessing change over time) | Baseline,12 months, 24 months
  Neuropsychological assessment of motor skills
Verbal Fluency (Assessing change over time) | Baseline,12 months, 24 months
  Neuropsychological assessment of language and communication skills
Demographic Information | Baseline
  Demographic data about the participant
Client Service Receipt Inventory (CSRI) Assessing change over time | Baseline, 12 months, 24 months
  Economic measure of health service use including frequency services are used (inc. mental health, physical health, criminal justice, council activities) and medication currently used (inc. measuring dosage, frequency, medication name, and how long its been taken for)
Schedule for Economic Data from Patient Records | Baseline, 12 months, 24 months
  Health information from patient notes to inform economic analysis
Questionnaire about the Process of Recovery (QPR) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Evaluates how participants view their recovery
Work Productivity and Activity Questionnaire (WPAI) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Measure of the effect of health problems on occupational functioning (i.e. ability to work and perform normal daily activities)
Relapse Questionnaire (Assessing change over time) | 6 months, 12 months, 24 months
  Self-report measure of any recent experience of what the patient or their close ones would describe as a relapse (severe or non-severe). Developed for this trial to identify instances of severe and non-severe relapse.
Medication Adherence Rating Scale (MARS-5) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Self-report measure of how participant is currently using antipsychotic medication (medication adherence)
Client Satisfaction Questionnaire (CSQ 8) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Patient satisfaction with mental health services.
EQ-5D-5L (Euroqol five levels- Assessing change over time) | Baseline, 6 months, 12 months, 24 months
  Measure of health status
ICECAP-A (ICEpop CAPability measure for Adults) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Measure of quality of life
Arizona Sexual Experiences Scale (ASEX) Assessing change over time | Baseline, 6 months, 12 months, 24 months
  Evaluates sexual functioning

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Moncrieff, MBBS, Principal Investigator — NHS / UCL
Locations (1):
- University College London, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moncrieff J, Crellin N, Stansfeld J, Cooper R, Marston L, Freemantle N, Lewis G, Hunter R, Johnson S, Barnes T, Morant N, Pinfold V, Smith R, Kent L, Darton K, Long M, Horowitz M, Horne R, Vickerstaff V, Jha M, Priebe S. Antipsychotic dose reduction and discontinuation versus maintenance treatment in people with schizophrenia and other recurrent psychotic disorders in England (the RADAR trial): an open, parallel-group, randomised controlled trial. Lancet Psychiatry. 2023 Nov;10(11):848-859. doi: 10.1016/S2215-0366(23)00258-4. Epub 2023 Sep 28. PMID 37778356
- See also: RADAR website — http://www.ucl.ac.uk/psychiatry/antipsychotic-discontinuation-and-reduction